CLINICAL TRIAL: NCT03030833
Title: Dysfunctional Hemoglobin Pulse Oximeter
Brief Title: Dysfunctional Hemoglobin Pulse Oximetry
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: QATP3040
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-01

CONDITIONS: Carbon Monoxide Poisoning
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Pulse Oximeter — Comparison of pulse oximetry to blood gas analyzer.

SUMMARY:
The purpose of the study is to assess device performance in the presence of carbon monoxide.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female.
* The subject is of any racial or ethnic group.
* The subject is between 18 years and 50 years of age (self-reported).
* The subject does not have significant medical problems (self-reported).
* The subject is willing to provide written informed consent and is willing and able to comply with study procedures.
* Exclusion Criteria:
* Has a BMI greater than 30.0 (calculated from self-reported weight and height).
* Has had any relevant injury at the sensor location site (self-reported).
* Has a deformity or abnormalities that may prevent proper application of the device under test (based on visual inspection).
* Has a known respiratory condition (self-reported).
* Is currently a smoker (self-reported).
* Has a known heart or cardiovascular condition (self-reported).
* Is currently pregnant (positive serum pregnancy test at screening visit or positive urine POC test on day of study).
* Is female and actively trying to get pregnant (self-reported).
* Has a clotting disorder (self-reported).
* Has Raynaud's Disease (self-reported).
* Is known to have anemia (hemoglobin value below lower range of normal for gender)
* Is known to have a hemoglobinopathy such as sickle-cell anemia or thalassemia (abnormal hemoglobin electrophoresis).
* Is known to have a inherited or congenital methemoglobinemia (self-reported).
* Has unacceptable collateral circulation from the ulnar artery (based on exam).
* Is unwilling or unable to provide written informed consent to participate in the study.
* Has another health condition which in the opinion of the principal investigator makes him/her unsuitable for testing.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Healthy male and females.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Carboxyhemoglobin accuracy | Through study completion, an average of 3 months.
  Values from the test device will be compared to the values from co-oximetry to determine accuracy of the test device.

CONTACTS AND LOCATIONS:
Overall Officials: David B MacLeod, MD, Principal Investigator — Duke University
Locations (1):
- HPPL Duke Univeristy, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No